CLINICAL TRIAL: NCT00514917
Title: A Randomized, Open Label, Multicenter, Phase III, 2-Arm Study of Androgen Deprivation With Leuprolide, +/- Docetaxel for Clinically Asymptomatic Prostate Cancer Subjects With a Rising PSA Following Definitive Local Therapy
Brief Title: A Study of Androgen Deprivation With Leuprolide, +/- Docetaxel for Clinically Asymptomatic Prostate Cancer Participants With a Rising Prostate Specific Antigen (PSA)
Acronym: Rising PSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision to discontinue the study, not due to any safety or efficacy concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_3503; 2007-000323-17 (EudraCT Number)
Record Dates: First submitted 2007-08-02; First posted 2007-08-10 (Estimated); Results first posted 2013-11-04 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-08

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Leuprolide; luprolide acetate gel depot; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel+Leuprolide+Bicalutamide (Experimental): Participants received docetaxel 75 milligram per square meter (mg/m^2) intravenous infusion over 1 hour every 3 weeks up to 10 cycles (3 week cycle) along with leuprolide 22.5 mg injection subcutaneously every 12 weeks up to 18 months and bicalutamide 50 mg tablet orally once daily for first 4 weeks of treatment.
  Interventions: Drug: Docetaxel; Drug: Leuprolide; Drug: Bicalutamide
- Leuprolide+Bicalutamide (Active Comparator): Participants received leuprolide 22.5 mg injection subcutaneously every 12 weeks up to 18 months and bicalutamide 50 mg tablet orally once daily for first 4 weeks of treatment.
  Interventions: Drug: Leuprolide; Drug: Bicalutamide

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m^2 intravenous infusion over 1 hour every 3 weeks up to 10 cycles.
  Other Names: TAXOTERE®; XRP6976
  Arms: Docetaxel+Leuprolide+Bicalutamide
Drug: Leuprolide — 22.5 mg injection subcutaneously every 12 weeks up to 18 months.
  Other Names: Eligard®
Drug: Bicalutamide — 50 mg tablet orally once daily for first 4 weeks of treatment.

SUMMARY:
The primary objective was to evaluate and compare the efficacy of androgen deprivation with or without docetaxel as determined by the median progression free survival (PFS) over the period of 18-month therapy and at least 18-month follow-up.

The secondary objectives were:

* To assess cancer specific survival;
* To compare overall survival between the 2 treatment groups;
* To evaluate patient-reported outcomes including quality of life, fatigue, and sexual functioning as measured by 3 different assessments.

DETAILED DESCRIPTION:
The duration of the study per participant was to be at least 36 months, of which the treatment period was 18 months for all participants, followed by at least 18 months follow-up period.

Participants received study treatment for up to 18 months from the time of study therapy initiation or less if one of the following occurred: disease progression, unacceptable toxicity, death, participant refusal or treatment delay beyond the time frame that is permitted for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prostate adenocarcinoma pathologically confirmed
* History of radical prostatectomy (pre-operative radiation therapy to the prostate or pelvis or salvage radiation after radical prostatectomy was allowed)
* Demonstration of biochemical progression of disease based on prostate specific antigen (PSA) doubling time. The minimum PSA value for eligibility was greater than or equal to (>=) 1. PSA doubling time over three values must be equal to (=) 9 months with a minimum of 3 weeks between assessments
* Serum testosterone >=100 nanogram per deciliter (ng/dL)
* Karnofsky performance status (KPS) >=70 percent (%)
* Adequate organ function as defined by the following laboratory criteria:

  * White blood cells >=3500 per cubic millimeter (mm^3)
  * Absolute neutrophil count (ANC) >=1500 per mm^3
  * Platelet count >=100,000 per mm^3
  * Hemoglobin >= 10.0 gram per deciliter (g/dL)
  * Total Bilirubin less than or equal to (<=) upper limit of normal (ULN) unless due to Gilbert's disease
  * Creatinine l <= 1.5 milligram per deciliter (mg/dL) or creatinine clearance >=60 cubic centimeters per minute
  * Aspartate transaminase (AST), alanine transaminase (ALT) and alkaline phosphatase within pre-defined ranges
* Previous hormonal therapy was allowed provided that the total duration of therapy did not exceed 6 months
* Man of childbearing potential who was willing to consent to use effective contraception while on treatment and for at least 3 months thereafter
* Participant who was willing and was able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Clinically significant cardiac disease (New York Heart Association Class III/IV), or severe debilitating pulmonary disease
* Uncontrolled serious active infection
* Anticipated duration of life < 2 years
* Less than 5-year history of successful treatment for other cancers or concurrent active nonprostate cancer other than nonmelanoma dermatologic tumor
* Peripheral neuropathy >=Grade 2
* History of hypersensitivity reaction to Docetaxel or other drugs formulated with polysorbate 80, leuprolide, or bicalutamide
* Prior chemotherapy within the past 10 years (except non-taxane based chemotherapy for treatment of other cancers); concurrent treatment on another clinical trial or with any other cancer therapy including chemotherapy, immunotherapy, radiotherapy (except salvage radiation therapy), chemoembolization therapy, cryotherapy
* Other severe acute or chronic medical conditions including psychiatric disease, or significant laboratory abnormality requiring further investigation that may cause undue risk for the participant's safety, delay or prohibit protocol participation, or interfere with the interpretation of study results, and in the judgment of the investigator would make the participant inappropriate for entry into this study
* Radiographic findings suspicious for metastatic disease in the treating physician's clinical judgment. Participant who had radiographically suspicious pelvic lymph nodes prior to radial prostatectomy, but who, at the time of enrollment did not have suspicious adenopathy was eligible. Participant was eligible even if he/she had tumor-containing pelvic adenopathy at the time of surgery as long as at the time of enrollment there was no radiographically evident nodal disease in the clinician's opinion
* Participant was the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
* Participant unlikely to comply with protocol or research tests, for example, uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study
* Participant who participated in another clinical study/received investigational product within 30 days of screening

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2007-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barrett Childs, MD, Study Director — Sanofi
Locations (9):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Vilnius, Lithuania
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 53 sites in North America (the United States of America and Canada) and Europe. Study was terminated after all participants had completed treatment with docetaxel, but before all participants had completed 18 months follow-up. The termination was not due to any safety or efficacy concerns.
Period: Overall Study
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Started | 207 | 206
Treated | 196 | 204
Completed Study Treatment | 170 | 182
Testosterone-Specific Evaluable | 122 | 124
Completed | 81 | 91
Not Completed | 126 | 115
Not completed — Death | 4 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 18 | 16
Not completed — Discontinued due to study closure | 88 | 81
Not completed — Undefined | 11 | 5

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least part of one dose of any of the study drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide | Total
Number analyzed (Participants) | 196 | 204 | 400
Age Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.97) | 64.0 (6.97) | 64.6 (6.99)
Age, Customized [Number; unit: participants]
  Less Than (<) 65 Years | 86 (43.9) | 104 (51.0) | 190
  Greater Than or Equal to (>=) 65 to < 75 Years | 95 (48.5) | 89 (43.6) | 184
  >= 75 Years | 15 (7.7) | 11 (5.4) | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 196 | 204 | 400
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 175 | 184 | 359
  Black | 16 | 13 | 29
  Asian/Oriental | 1 | 0 | 1
  Others | 4 | 7 | 11
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meter (m^2)] — BSA was calculated using the Dubois and Dubois formula: BSA (in square meter) = (weight^0.425* height^0.725)*0.007184; where weight is in kilogram (kg) and height is in centimeter (cm). Here "N" (number of participants analyzed) = 192, 198 for each treatment arm, respectively.
  square meter (m^2) | 2.05 (0.176) | 2.08 (0.194) | 2.06 (0.186)
Prior Radiation Therapy [Number; unit: participants] | 63 | 75 | 138

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-Free Survival (PFS) in Intent-to-treat (ITT) Population
Description: PFS was the time from randomization to the date of first documented prostate specific antigen (PSA) progression, or radiographic progression, or death due to prostate cancer in the absence of previous documentation of disease progression, whichever occurred first. PSA progression was determined as: a) During treatment period: a 50 percent (%) increase from baseline, which was confirmed by a second value; b) During follow-up: detectable PSA (defined as PSA greater than or equal to 0.05 nanogram per millimeter [ng/mL]), which was confirmed by consecutive observation (not less than 2 weeks apart). Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Randomization until PSA progression or radiographic progression or death due to prostate cancer, assessed up to Month 60
Population: ITT population included all participants who were randomized, with study drug assignment designated according to randomization, regardless of whether participants received any study drug or a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 207 | 206
months | 25.4 [23.8 to 27.8] | 23.3 [22.6 to 25.1]
Statistical Analysis 1: Comparison: Docetaxel+Leuprolide+Bicalutamide vs Leuprolide+Bicalutamide; Null hypothesis: No difference between new treatment combination (Docetaxel+Leuprolide+Bicalutamide) and conventional treatment (Leuprolide+Bicalutamide). The study was sized to have 90% power to detect a difference between treatment arms at a 2-sided 0.05 significance level with 186 events and anticipating 10% non-evaluable participants; Test type: Superiority or Other; p = 0.0501, Log Rank — A priori threshold for statistical significance = 0.05; P-value was not adjusted for multiplicity of tests; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [1.00 to 1.65] — The hazard ratio Leuprolide+Bicalutamide vs. Docetaxel+Leuprolide+Bicalutamide was estimated using an un-stratified Cox proportional hazards model. A hazard ratio >1 indicates a lower risk of Docetaxel+Leuprolide, compared to Leuprolide

2. Primary Outcome: Progression-Free Survival (PFS) Rate at Month 36 in ITT Population
Description: PFS rate at Month 36 was defined as probability of being progression-free at Month 36. PFS rate was estimated using the Kaplan-Meier method.
Time Frame: Month 36
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percent chance of being progression-free
Groups:
- Docetaxel+Leuprolide+Bicalutamide: Participants received docetaxel 75 milligram per square meter (mg/m^2) intravenous infusion over 1 hour every 3 weeks up to 10 cycles along with leuprolide 22.5 mg/m^2subcutaneous injection for every 12 weeks up to 18 months and bicalutamide 50 mg tablet orally once daily for first 4 weeks of treatment.
- Leuprolide+Bicalutamide: Participants received leuprolide 22.5 mg/m^2 subcutaneous injection for every 12 weeks up to 18 months and bicalutamide 50 mg tablet orally once daily for first 4 weeks of treatment.
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 207 | 206
percent chance of being progression-free | 15.5 [9.1 to 23.3] | 8.6 [3.8 to 16.0]

3. Secondary Outcome: Overall Survival (OS): Number of Participants Who Died (All Cause)
Description: The OS was the time interval from the date of randomization to the date of death due to any cause. OS was to be analyzed using the Kaplan-Meier method. However, the analysis was not performed due to insufficient number of events. Reported is the number of participants who died from any cause.
Time Frame: Randomization until death due to any cause, assessed up to Month 60
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 207 | 206
participants | 4 | 11

4. Secondary Outcome: Cancer-Specific Survival: Number of Participants Who Died (Cancer-Specific)
Description: The cancer-specific survival was the time from the date of randomization to the date of death due to prostate cancer. Cancer-specific survival was to be analyzed using the Kaplan-Meier method. However, the analysis was not performed due to insufficient number of events. Reported is the number of participants who died from prostate cancer.
Time Frame: Randomization until death due to prostate cancer, assessed up to Month 60
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 207 | 206
participants | 2 | 3

5. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Total Score at End of Treatment (EOT)
Description: FACT-P is a 39-item participant questionnaire which assesses physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items), functional well-being (7 items), and additional prostate cancer specific concerns (12 items). All items are scored from 0 (not at all) to 4 (very much). The total FACT-P score ranges from 0-156, with higher scores representing a better quality of life with fewer symptoms. A score of 156 represents the best outcome.
Time Frame: Baseline, EOT (up to Month 18)
Population: ITT population. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure and "n" signifies participants evaluable at each time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 206 | 205
units on a scale
  Baseline (n=206, 205) | 121.4 (18.32) | 119.6 (17.95)
  Change at EOT (n=186, 184) | -4.9 (13.55) | -3.4 (14.78)

6. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Prostate (FACT-P) Trial Outcome Index (TOI) Score at EOT
Description: Physical well-being, functional well-being, and prostate cancer concerns sub-scales of the FACT-P questionnaire were combined to calculate TOI. Total TOI score ranges from 0 to 104, with higher scores representing a better quality of life with fewer symptoms.
Time Frame: Baseline, EOT (up to Month 18)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 206 | 206
units on a scale
  Baseline (n=206, 206) | 82.1 (12.58) | 80.4 (12.52)
  Change at EOT (n=187, 187) | -5.4 (10.19) | -3.1 (11.83)

7. Primary Outcome: Median Progression-Free Survival (PFS) in Testosterone Specific Evaluable Population
Description: PFS was the time from randomization to the date of first documented PSA progression, or radiographic progression, or death due to prostate cancer in the absence of previous documentation of disease progression, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: Testosterone-specific evaluable population included all participants who recovered testosterone to non-castrate levels (50 ng/mL) following the completion of treatment of leuprolide with at least 1 follow-up PSA assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 122 | 124
months | 25.7 [25.1 to 28.1] | 24.7 [22.8 to 25.3]

8. Secondary Outcome: Change From Baseline in Multidimensional Assessment of Fatigue (MAF) Index Score at EOT
Description: MAF scale consists of 16-items to measure 4 dimensions of fatigue during past week: severity (Item 1-2), distress (Item 3), degree of interference in activities of daily living (Item 4-14), and timing (Item 15-16). Item 1-14 are scored on a numeric rating scale from 1 to 10, where higher score indicate more severity/distress/interference. Item 15-16 had multiple choice responses (4 responses each). Scale Index was calculated using Item 1-15, in following steps: 1) Item 15 score converted to 1-10 scale by multiplying the score with 2.5; 2) Average score was calculated from Item 4-14; 3) Finally scale index was calculated by adding Items 1, 2, 3 scores with average score from step 2 and converted score of Item 15 from step 1. Total MAF scale index score ranges 1 (no fatigue) to 50 (severe fatigue).
Time Frame: Baseline, EOT (up to Month 18)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 168 | 171
units on a scale
  Baseline (n=168, 171) | 16.4 (7.33) | 16.6 (7.93)
  Change at EOT (n=127, 144) | 4.0 (8.93) | 2.6 (8.60)

9. Primary Outcome: Progression-Free Survival (PFS) Rate at Month 36 in Testosterone Specific Evaluable Population
Description: as for outcome 2
Time Frame: Month 36
Population: Testosterone-specific evaluable population included all participants who recovered testosterone to non-castrate levels (50 ng/mL) following completion of treatment of leuprolide with at least 1 follow-up PSA assessment.
Measure: Number (95% Confidence Interval); unit: percent chance of being progression-free
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 122 | 124
percent chance of being progression-free | 15.8 [9.0 to 24.3] | 9.1 [4.0 to 16.7]

10. Secondary Outcome: Change From Baseline in Erectile Function Domain of International Index of Erectile Function (EF-IIEF) Total Score at EOT
Description: EF-IIEF is a 6-item erectile function domain of IIEF. It consists of Question 1, 2, 3, 4, 5, and 15 of IIEF questionnaire. 5 questions are scored from 0 (no activity) to 5 (very high activity) and 1 question is scored from 1 (very low activity) to 5 (very high activity). Total EF-IIEF score ranges from 1 to 30, where higher score indicates high activity.
Time Frame: Baseline, EOT (up to Month 18)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 201 | 205
units on a scale
  Baseline (n=201, 205) | 6.4 (8.30) | 6.8 (8.25)
  Change at EOT (n=180, 186) | -3.1 (7.15) | -3.3 (7.11)

11. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAE: any adverse event (AE) that occurred or worsened during the on-treatment period, which was the period from first administration of study treatment until 30 days after last administration of study treatment. AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly, or medically important. Drug-related AEs were any untoward medical occurrences attributed to study drug in a participant who received study drug. National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 Grade 3 (severe) and Grade 4 (life threatening/disabling) TEAEs were also reported.
Time Frame: From first administration of study treatment until 30 days after the last administration of study treatment
Population: Safety population included all randomized participants who received at least part of one dose of any of the study drugs.
Measure: Number; unit: participants
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Number analyzed (Participants) | 196 | 204
participants
  Any TEAE | 188 | 163
  Any Serious AE | 49 | 20
  Any TEAE Resulting in Death | 0 | 1
  Any TEAE Leading to any Treatment Discontinuation | 35 | 1
  Any Grade 3-4 TEAE | 94 | 22
  Docetaxel Related TEAE | 183 | NA — Participants in this treatment arm did not receive docetaxel.
  Leuprolide Related TEAE | 109 | 136
  Bicalutamide Related TEAE | 52 | 74
  Any Treatment Related TEAE | 184 | 136
  Any Grade 3-4 Serious TEAE | 43 | 14
  Any TEAE Leading to Interruption of any Treatment | 77 | 1

ADVERSE EVENTS:
Time Frame: From signature of the informed consent form up to the last visit in the study
Description: The analysis was performed on safety population, defined as all randomized participants who received at least part of one dose of any of the study drugs, and included all TEAEs that developed or worsened from first administration of study treatment until 30 days after last administration of study treatment.
Arm/Group | Docetaxel+Leuprolide+Bicalutamide | Leuprolide+Bicalutamide
Serious Adverse Events (participants affected / at risk) | 49/196 | 20/204
Other Adverse Events (participants affected / at risk) | 185/196 | 139/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel+Leuprolide+Bicalutamide (N=196) | Leuprolide+Bicalutamide (N=204)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 11 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 9 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 3 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 2
AORTIC VALVE DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
NODAL ARRHYTHMIA (Cardiac disorders) | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
RETINAL DETACHMENT (Eye disorders) | 0 | 1
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
PERITONITIS (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL WALL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
COLITIS (Gastrointestinal disorders) | 0 | 1
CHEST PAIN (General disorders) | 1 | 1
GENERALISED OEDEMA (General disorders) | 1 | 0
HERNIA (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
NON CARDIAC CHEST PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 1 | 0
ANAPHYLACTOID REACTION (Immune system disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0
GENITOURINARY TRACT INFECTION (Infections and infestations) | 1 | 0
NEUTROPENIC INFECTION (Infections and infestations) | 1 | 0
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS PERFORATED (Infections and infestations) | 0 | 1
BACTERAEMIA (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 0 | 1
GROIN ABSCESS (Infections and infestations) | 0 | 1
UROSEPSIS (Infections and infestations) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
DIZZINESS (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
MYASTHENIA GRAVIS (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel+Leuprolide+Bicalutamide (N=196) | Leuprolide+Bicalutamide (N=204)
NEUTROPENIA (Blood and lymphatic system disorders) | 31 | 0
ANAEMIA (Blood and lymphatic system disorders) | 18 | 2
LACRIMATION INCREASED (Eye disorders) | 31 | 0
DIARRHOEA (Gastrointestinal disorders) | 64 | 7
NAUSEA (Gastrointestinal disorders) | 56 | 11
CONSTIPATION (Gastrointestinal disorders) | 28 | 9
STOMATITIS (Gastrointestinal disorders) | 20 | 0
VOMITING (Gastrointestinal disorders) | 19 | 2
DYSPEPSIA (Gastrointestinal disorders) | 17 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 10 | 3
FATIGUE (General disorders) | 104 | 58
OEDEMA PERIPHERAL (General disorders) | 66 | 11
PYREXIA (General disorders) | 24 | 0
ASTHENIA (General disorders) | 19 | 3
NASOPHARYNGITIS (Infections and infestations) | 12 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 2
WEIGHT INCREASED (Investigations) | 13 | 13
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 12 | 7
WEIGHT DECREASED (Investigations) | 11 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 24 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 15 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 40 | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 34 | 12
MYALGIA (Musculoskeletal and connective tissue disorders) | 31 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 | 8
BONE PAIN (Musculoskeletal and connective tissue disorders) | 13 | 1
DYSGEUSIA (Nervous system disorders) | 51 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 37 | 3
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 31 | 4
HEADACHE (Nervous system disorders) | 21 | 10
PARAESTHESIA (Nervous system disorders) | 19 | 1
HYPOAESTHESIA (Nervous system disorders) | 16 | 3
DIZZINESS (Nervous system disorders) | 15 | 8
INSOMNIA (Psychiatric disorders) | 31 | 9
POLLAKIURIA (Renal and urinary disorders) | 15 | 7
URINARY INCONTINENCE (Renal and urinary disorders) | 12 | 17
COUGH (Respiratory, thoracic and mediastinal disorders) | 26 | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 25 | 11
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 14 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 12 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 110 | 3
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 50 | 1
RASH (Skin and subcutaneous tissue disorders) | 18 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 15 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 11 | 0
HOT FLUSH (Vascular disorders) | 82 | 118
HYPERTENSION (Vascular disorders) | 8 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall provide the Steering Committee a copy of any manuscript, abstract or oral communication derived from the study for review and comment at least 30 days in advance of any submission. The Sponsor's representatives shall have the right to review and/or delay any publication or presentation to prevent disclosure of Sponsor's confidential information and preserve intellectual property rights.